CLINICAL TRIAL: NCT02068079
Title: A Pilot Study of Trientine With Vemurafenib for the Treatment BRAF Mutated Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045015
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Trientine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib and Trientine (Other)
  Interventions: Drug: Vemurafenib and Trientine

INTERVENTIONS:
Drug: Vemurafenib and Trientine

SUMMARY:
The purpose of this study is to evaluate the safety of combination therapy with vemurafenib and trientine in patients with BRAF mutated metastatic melanoma.

Vemurafenib is a drug that is currently approved by the United States Food and Drug Administration (FDA) and by the European Medicines Agency (EMA) to treat adult patients with melanoma that has spread to other parts of the body or cannot be removed by surgery. It can only be used in patients whose cancer has a change (mutation) in the "BRAF" gene.

Preclinical data suggests that use of a copper chelator (reducer) is a strategy to block cellular signaling activity which would result in anti-tumor effects (slow tumor growth). Trientine is a copper chelator and is FDA approved for the treatment of Wilson's disease (a disease of copper metabolism) and is generally well tolerated. It works by binding to copper to help remove it from the body. Trientine is not FDA approved for the treatment of melanoma and its use in this study is investigational. "Investigational" means the study drug is still being tested in research studies.

All patients will receive vemurafenib at 960mg PO twice daily with continuous dosing in combination with trientine in escalating doses. The dose of trientine will depend on what portion of the study.

In order to participate in the study, patients must test positive for the change (mutation) in the BRAF gene.

ELIGIBILITY:
Inclusion criteria

1. Willing and able to give written informed consent.
2. ECOG performance status ≤ 1
3. Histologic diagnosis of unresectable stage IIIC or stage IV melanoma that is BRAF V600 mutation positive
4. Stable, treated brain metastases are allowed. Stable brain metastases are defined as stable on MRI 4 weeks after the completion of radiation, and currently asymptomatic no longer requiring corticosteroids for 2 weeks prior to the initiation of study drug.
5. Cutaneous tumor deposits that, in the opinion of the investigator are amenable to sequential biopsies for correlative analyses. In addition to these, all patients must have measurable disease (i.e., present with at least one measurable lesion per RECIST, version 1.1).
6. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
7. Required values for initial laboratory tests:

   * WBC ≥ 2000/uL
   * ANC ≥ 1000/uL
   * Platelets ≥ 75 x 103/uL
   * Hemoglobin ≥ 9 g/dL (≥ 80 g/L; may be transfused)
   * Creatinine ≤ 2.0 x ULN
   * AST/ALT ≤ 2.5 x ULN for patients without liver metastasis, ≤ 5 times for liver metastases
   * Bilirubin ≤ 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

   * Amenorrhea ≥ 12 consecutive months without another cause, or
   * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours.

Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria

1. Prior treatment with a BRAF or MEK inhibitor for metastatic melanoma (treatment in the adjuvant setting is allowed)
2. Any other malignancy form which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or DCIS. Patients with prior malignancies that are not considered to be an active problem may be enrolled at the discretion of the investigator, regardless of time frame.
3. Women of childbearing potential (WOCBP), defined above in Section 4.1, who:

   1. are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
   2. have a positive pregnancy test at baseline, or
   3. are pregnant or breastfeeding.
4. Anti-cancer therapy within 28 days prior to starting on therapy
5. Any serious or unstable pre-existing medical conditions psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
6. Known history of Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed).
7. A history or evidence of cardiovascular risk including any of the following:

   1. A QTc interval ≥ 500 ms at screening
   2. A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with atrial fibrillation controlled for > 30 days prior to randomization are eligible.
   3. A history (within 6 months prior to randomization) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty
   4. A history or evidence of current ≥Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines
   5. Treatment refractory hypertension defined as a blood pressure of systolic> 150 mmHg and/or diastolic > 100 mm Hg which cannot be controlled by antihypertensive therapy;
   6. Patients with intra-cardiac defibrillators or permanent pacemakers;
8. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

   a. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes)
9. Females who are nursing
10. A known diagnosis of Wilson's disease.
11. Patients with clinical symptoms consistent with active gastritis.
12. Patients with a condition that, in the opinion of the investigator, would interfere with the absorption of oral medication will be excluded from the study.
13. Patients requiring iron supplementation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 Cycle (4 Weeks)
  Maximum Tolerated Dose is defined as the highest dose level in which ≤1 of 6 patients experience a dose limiting toxicity.

SECONDARY OUTCOMES:
Overall Response | 1 year
  The number of complete and partial responses using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee v 1.1
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from study enrollment to disease progression or death due to any cause, whichever comes first.
Overall Survival (OS) | 2 years
  OS is defined from enrollment to death due to any cause.
The change in phosphorylated Erk kinase activity relative to total Erk kinase activity | Pre-treatment; two weeks into combination therapy (day 15), and at the time of disease progression while still on combination therapy, up to 2 years
The change in phosphorylated MEK kinase activity relative to total MEK kinase activity | Pre-treatment; two weeks into combination therapy (day 15), and at the time of disease progression while still on combination therapy, up to 2 years
The change in the expression of the copper transporter CTR1 | Up to 2 years
  Change will be measured as the percent change compared to the baseline status
Incidence of hyperproliferative skin lesions, specifically cutaneous squamous cell carcinomas and keratoacanthomas | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: April K Salama, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States